CLINICAL TRIAL: NCT01317693
Title: Extracorporeal Shock Wave Therapy With a Wide Focus Probe for the Treatment of Erectile Dysfunction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, i_gruenwald, MD, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0571-10-RMB
Record Dates: First submitted 2011-03-08; First posted 2011-03-17 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Erectile Dysfunction
Keywords: LI-ESWT; Erectile Dysfunction; ED; Shock waves; Therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment LI-ESWT (Experimental): Device: Extracorporeal Shockwave Therapy Generator (Omnispec model ED1000) Gel is spread around the penis and on the Shock Wave applicator and Treatment (12 sessions in total) of 300 shocks per site, on 5 penile anatomical sites.
  Interventions: Device: Low intensity shock waves

INTERVENTIONS:
Device: Low intensity shock waves — 1500 shocks, Energy Density - 0.09 mJ/mm2
  Other Names: Omnispec model ED1000

SUMMARY:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to the penile tissue. Shockwaves are created by a special generator and are focused using a specially designed shockwave applicator apparatus. The shockwaves are delivered through the applicator covering the corpora cavernosa of the penis. In previous studies the investigators used a medium focused probe and in this study the investigators are evaluating results of this therapy using a wider focus probe in the aim of improving results of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* At least 50% unsuccessful to attempt sexual intercourse for 4 times at 4 different days
* Positive response to PDE-5 inhibitors
* IIEF-5 domain score of 12-20 denoting mild to severe ED
* Non-Neurological pathology
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* NPT - normal/flat
* Prior prostatectomy surgery
* Any cause of ED other than vascular related
* Any unstable medical, psychiatric, spinal cord injury, penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Cardiovascular conditions that prevent sexual activity
* History of heart attack, stroke or life-threatening arrhythmia within the prior 6 months.
* Cancer within the past 5 years.
* Anti-androgens, oral or injectable androgens
* Use of any treatment for ED within 7 days of screening including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in IIEF-ED Domain Questionaire Score > 5 points is considered treatment success | 13 weeks

SECONDARY OUTCOMES:
Rigidity Score Questionaire- an increase by at least 1 point is considered success | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Rambam Health Care Campus; Yoram Vardi, Prof., Study Director — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel